CLINICAL TRIAL: NCT05415332
Title: The Current Status and Clinical OUTcomes of Cardiogenic Shock Patients And the Role of Specialist in Cardiovascular Critical Care Unit
Acronym: SCOUT SPARC
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-0383
Record Dates: First submitted 2022-06-01; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiogenic shock patients: We will collect patient's demographic information, medical history, vital signs, cardiac arrest, the maximum dose of the drug at shock treatment and whether mechanical circulatory support devices are inserted, indicators of deterioration and improvement of shock.
  For follow-up observations, only prospective subjects are examined for results and administrative information conducted by visiting an outpatient at the time of one, six, one, two, three, four, and five or more years after the shock.
- Patients hospitalized in cardiovascular intensive care unit: we will collect patient's demographic information, medical history related to cardiovascular disease, and vital signs on the admission date to the cardiovascular critical care unit.

SUMMARY:
In the case of cardiogenic shock, the early mortality rate is the highest compared to other types of shock, but it is characterized by a good prognosis and quality of life after recovery, so monitoring the treatment progress is very important to identify the patient's prognosis. However, there are few studies specifically reported on hemodynamic monitoring and prognosis of cardiogenic shock. In addition, as mechanical circulatory support devices are in the spotlight, studies on their effects and safety are starting, but studies on cardiogenic shock are often limited to patients with myocardial infarction.

This study is a prospective and retrospective cohort observational study, we aim to identify factors that can improve prognosis, including various drug treatments, diagnostic techniques, and mechanical circulatory support device by investigating the treatment status and clinical outcomes of patients with cardiogenic shock hospitalized in cardiovascular critical care unit. In addition, the purpose of this study is to investigate the association between the prognosis of patients with cardiogenic shock and the presence of a specialist resident during regular work hours to clarify the role and necessity of a resident specialist in the cardiovascular intensive care unit.

Furthermore, by predicting and treating the clinical course of patients with cardiogenic shock at an early stage, the aim is to reduce the mortality rate and improve the patients' ability to perform daily activities.

ELIGIBILITY:
Inclusion Criteria:

(prospective)

1. Patients over 19-year-old
2. Patients who are hospitalized in the cardiovascular critical care unit for cardiogenic shock or reduced blood pressure due to other causes.

   2-1) In the event that the systolic blood pressure is less than 90mmHg for at least 30 minutes despite fluid treatment, or the use of vasopressor drug is required to maintain systolic blood pressure more than 90mmHg.

   2-2) patients have at least one of the symptoms of peripheral tissue hypoperfusion (cold skin, urineoutput < 30cc/ hour, decreased consciousness, lactate > 2.0mmol/l) or pulmonary edema.

   2-3) Patients supported by Mechanical Circulatory support device
3. Where the cause of a cardiogenic shock conforms to one or more of the following matters:

   3-1) In the case of an intervention or surgery has been performed due to coronary artery disease, peripheral artery disease, venous thromboembolism, pulmonary artery disease, aortic disease, etc.

   3-2) In the case of an intervention or surgery has been performed due to valve disease.

   3-3) In the case of the insertion of an instrument in the heart is performed due to atrial defect, left atrium, arteriosclerosis, etc.

   3-4) In the case of ablation or surgery, defibrillator implantation, and pacemaker implantation.

   3-5) In the case of pericardiocentesis or window formation has been performed due to cardiac tamponade.

   3-6) When monitoring is required for hypothermia therapy after spontaneous circulation recovery.

   3-7) When monitoring is required after other heart-related procedures or surgery 3-8) When monitoring is required after heart transplant
4. Where a patient or legal representative voluntarily agrees to access medical records and data necessary for this study during the entire study period

(retrospective) Patients over 19-year-old who treated in the cardiovascular critical care unit from January 1, 2018 to the IRB approval date for decreased blood pressure or needed intensive monitoring of vital signs.

Exclusion Criteria:

1. A patient with irreparable brain damage.
2. If there are no witnesses outside the hospital during cardiac arrest.
3. DNR(Do Not Resuscitate) patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (prospective) Patients over 19-year-old who have been hospitalized in cardiovascular critical care unit for cardiogenic shock and other causes of decreased blood pressure after the IRB approval date.
  (retrospective) Patients over 19-year-old who treated in the cardiovascular critical care unit from January 1, 2018 to the IRB approval date for decreased blood pressure or needed intensive monitoring of vital signs.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
In-hospital death | 30 days after onset of cardiogenic shock
  Death during hospitlization

SECONDARY OUTCOMES:
In-hospital cardiac death | 30 days after onset of cardiogenic shock
  cardiac death during hospitlization
Defective neurological indicators | 30 days after onset of cardiogenic shock
  Measurement using CPC(Cerebral perfomance category) score
cardiac death within 30 days | 30 days after onset of cardiogenic shock
  30 Days mortality
all cause of death within 30 days | 30 days after onset of cardiogenic shock
  30 Days mortality
all cause of death during follow-up | Outpatient visits at the time of one month, six months, one year, two years, three years, four years and five years from the date of the cardiogenic shock.
  all cause of death during follow-up
Major Adverse Cardiovascular Events during follow-up | Outpatient visits at the time of one month, six months, one year, two years, three years, four years and five years from the date of the cardiogenic shock.
  Major Adverse Cardiovascular events(MACE) is defined CVD events, admission for heart failure, ischemic cardiovascular events, bleeding events, cardiac death, heart transplactation, other thromboembolism
successful weaning of mechanical circulatory support device | 30 days after onset of cardiogenic shock
  if successful weaning of mechanical circulatory support device or not

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Min Ahn, Principal Investigator — Yonsei University Health system Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No